CLINICAL TRIAL: NCT06587568
Title: Mobile Chat Messaging Plus Screening-based Brief Alcohol Intervention for Patients With Chronic Liver Diseases: a Pilot Randomised Controlled Trial
Brief Title: Mobile Chat Messaging for Alcohol Reduction in Patients With Chronic Liver Diseases
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Health and Medical Research Fund (Other Government)
Responsible Party: Principal Investigator, Tzu Tsun Luk, Research Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21222731
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Chronic Liver Disease
Keywords: drinking; cirrhosis; hepatitis; SBIRT; WhatsApp; Chinese; mHealth; ABI
MeSH Terms: conditions — Fibrosis; Hepatitis | interventions — Mass Screening; Crisis Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mobile chat messaging (Experimental): Mobile chat messaging + Screening-based alcohol intervention
  Interventions: Behavioral: Mobile chat messaging; Behavioral: Screening, brief intervention and referral to treatment
- Brief intervention (Active Comparator): Screening-based alcohol intervention only
  Interventions: Behavioral: Screening, brief intervention and referral to treatment

INTERVENTIONS:
Behavioral: Mobile chat messaging — A trained counsellor will interact with a participant individually and provide personalised alcohol reduction information and advice via a mobile instant messaging app in real time for 3 months from randomisation.
  Arms: Mobile chat messaging
Behavioral: Screening, brief intervention and referral to treatment — Brief counselling (5 to 10 mins) to reduce drinking and a self-help booklet
  Other Names: SBIRT

SUMMARY:
The goal of this pilot randomized controlled trial is to evaluate the trial feasibility and acceptability of mobile chat messaging for reducing alcohol use among patients with chronic liver diseases. Specific objectives include:

1. To assess whether the eligibility criteria were too restrictive by estimating the eligibility rate
2. To assess how many eligible CLD patients accepted the invitation to participate in the trial
3. To assess the participant retention rate through 6 months after treatment initiation
4. To assess the intervention acceptability in terms of participants' engagement with and rating of the chat messaging intervention.
5. To assess the safety of the intervention
6. To estimate the intervention effect on alcohol use outcomes and liver functions
7. To synthesise data to inform the sample size calculation in the future definitive trial
8. To explore the participants' perception and experiences in the chat-based intervention

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Diagnosed with chronic liver disease
3. Alcohol Use Disorders Identification Test score ≥8
4. Own a smartphone with a mobile instant messaging app installed
5. Able to read and communicate in Chinese

Exclusion Criteria:

1. Having a psychiatric or psychological disease or on psychotropic drugs
2. Participating in other alcohol reduction or abstinence programmes
3. Require emergency or in-patient treatment after consultation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2024-10-02 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | Through recruitment completion, about 8 months
  Number of participants divided by the number of eligible subjects
Retention rate | 6 months after randomisation
  Number of participants completed the follow-up divided by the number of participants
Weekly alcohol consumption | 6 months after randomisation
  Assessed by questions 1 and 2 of AUDIT-C

SECONDARY OUTCOMES:
Eligibility rate | Through recruitment completion, about 8 months
  Number of eligible patients divided by the number of patients screened
Weekly alcohol consumption | 3 months after randomisation
  Assessed by questions 1 and 2 of AUDIT-C
Frequency of heavy episodic drinking | 3 months after randomisation
  Self-reported
Frequency of heavy episodic drinking | 6 months after randomisation
  Assessed by question three of AUDIT-C
AUDIT score and level | 3 months after randomisation
  Assessed by the Alcohol Use Disorders Identification Test
AUDIT score and level | 6 months after randomisation
  Assessed by the Alcohol Use Disorders Identification Test
Total alcohol consumption in the past week | 6 months after randomisation
Past 7-day alcohol abstinence | 3 months after randomisation
  Self-reported
Past 7-day alcohol abstinence | 6 months after randomisation
  Self-reported
Past 30-day alcohol abstinence | 3 months after randomisation
  Self-reported
Past 30-day alcohol abstinence | 6 months after randomisation
  Self-reported
Past 7-day total alcohol consumption | 3 months after randomisation
  Measured in grams

CONTACTS AND LOCATIONS:
Overall Officials: Tzu Tsun Luk, PhD, RN, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided